CLINICAL TRIAL: NCT04224259
Title: Utility of Vertical Puncture Technique Assisted by Ultrasound Pre-scan to Reduce Needle Redirection During Right Jugular Vein Cannulation
Brief Title: Ultrasound Pre-scan to Reduce Needle Redirection During Right Jugular Vein Cannulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: N201803005
Record Dates: First submitted 2019-10-28; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia
Keywords: Ultrasound; pre-scan; right internal jugular vein

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound pre-scan group (Experimental): Perform ultrasound pre-scan before central venous cannulation
  Interventions: Procedure: Ultrasound pre-scan
- landmark guidance group (Sham Comparator): Use the traditional landmark method to perform central venous cannulation
  Interventions: Procedure: Landmark guidance

INTERVENTIONS:
Procedure: Ultrasound pre-scan — Before cannulation, use ultrasound to mark the position of right internal jugular vein
  Arms: ultrasound pre-scan group
Procedure: Landmark guidance — The traditional landmark-guided technique for internal jugular vein cannulation, including recognizing the sternocleidomastoid muscle and palpating the carotid artery
  Arms: landmark guidance group

SUMMARY:
This study aims to define a simple, safe, and effective ultrasound pre-scan technique for right internal jugular vein (RIJV) cannulation. After placing the patient properly, the operator puts a linear ultrasound probe at the mid neck in short-axis view. With the IVJ in the center of the screen, the operator makes marks at both ends of the transducer (mark A and B), and then rotates the transducer 90 degrees counterclockwise. After finding IJV in long-axis view with transducer vertical to the ground, other two marks are made at both ends of the transducer (mark C and D). After proper preparation, the operator recognizes the cross point made by the imagined lines of marks AB and marks CD (point E). The needle is inserted vertically to the ground at point E.

Inclusion criteria are adult patients receiving general anesthesia in need of central venous cannulation.The primary endpoint is the number of needle redirection, and secondary endpoints include first attempt success rate, artery puncture, complication, number of wire attempt, number of skin insertion, venous access time, catheterization time, and malposition. The hypothesis is that this ultrasound pre-scan method would have a fewer number of needle redirection, a higher first-attempt success rate, as well as less complication, number of redirection.

DETAILED DESCRIPTION:
Ultrasound-guided central venous cannulation has been widely used because of lower technical failure rate and complications, and faster access compared with landmark-guided cannulation. Real-time guidance is more complex to perform and time-consuming in comparison to pre-scan technique. Therefore, real-time guidance should be reserved to specific groups, such as infants, children, or those with anatomical abnormality. However, there's no widely accepted ultrasound pre-scan techniques yet. The aim of this study is to define a simple, safe, and effective ultrasound pre-scan technique for right internal jugular vein (RIJV) cannulation.

Patient position for RIJV cannulation was reviewed in detail. First, 15ﾟ Trendelenburg tilt significantly increases the diameter of right internal jugular vein. Second, extreme head rotation to the opposite side will increase the overlap percentage between IJV and common carotid artery (CCA), but neutral head position might make the procedure difficult. Neutral head position or small degree (≦15ﾟ) of head rotation was recommended. Third, although shoulder roll is not recommended since it decreases the anterior-posterior diameter of RIJV, 4- to 5cm-high shoulder roll could be used to reduce the overlap if needed10. In conclusion, patients should be positioned by a 15ﾟ Trendelenburg tilt and 15ﾟ head rotation to the opposite side without a shoulder roll unless the IJV is anterior to CCA, which was termed as the rule of 15 by the research team.

After placing the patient properly, the operator puts a linear ultrasound probe at the mid neck in short-axis view. With IVJ in the center of the screen, marks at both ends of the transducer (mark A and B) are made. Then the operator rotates transducer 90 degrees counterclockwise. After finding IJV in long-axis view with transducer vertical to the ground, other two marks are made at both ends of the transducer (mark C and D), and transducer and jelly are removed. Then the operator sterilizes the performing field with chlorhexidine without removing the marks. After proper preparation and recognizing the cross point made by the imagined lines of marks AB and marks CD (point E), the operator inserts the needle vertically to the ground at point E.

The aim of this study is to compare the effectiveness and safety between ultrasound pre-scan technique and traditional landmark-guidance. Inclusion criteria are adult patients receiving general anesthesia in need of central venous cannulation. The primary endpoint is the number of needle redirection, and secondary endpoints include first attempt success rate, artery puncture, complication, number of wire attempt, number of skin insertion, venous access time, catheterization time, and malposition. The hypothesis is that the ultrasound pre-scan method would have a fewer number of needle redirection, a higher first-attempt success rate, as well as less complication, number of redirection.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years and younger than 80 years of age
* American Society of Anesthesiologists Physical Status Classification I-III (no immediate life-threatening condition)
* Scheduled for regular surgery
* Receive general anesthesia with endotracheal tube intubation
* In need of central venous catheter placement

Exclusion Criteria:

* Body Mass Index > 35kg/m^2
* Abnormal anatomy of the neck
* Limited range of motion of the neck
* The surgery does not allow right internal jugular vein cannulation or other contraindications for the procedure

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
number of needle redirection | During the cannulation procedure
  How many times of the needle being withdrawn and redirected before successfully access internal jugular vein

SECONDARY OUTCOMES:
first attempt success rate | During the cannulation procedure
  successfully access the internal jugular vein at first attempt
artery puncture | During the cannulation procedure
  accidental artery puncture
number of wire attempt | During the cannulation procedure
  how many times of the wire attempts before successful wire insertion to internal jugular vein
number of skin insertion | During the cannulation procedure
  how many different skin insertion sites were tried before successfully access the internal jugular vein
venous access time | During the cannulation procedure
  How long does it take from the first skin insertion to success venous access
catheterization time | During the cannulation procedure
  How long does it take from the first skin insertion to successful catheter cannulation
malposition | During the cannulation procedure
  the catheter misplaced to wrong sites (e.g. artery, subcutaneous)
presence of hematoma | immediately at the end of procedure, evaluated by clinical signs and ultrasound image
  a different and blinded investigator reviewed the post-procedure ultrasound image to determine whether there is hematoma after the procedure
other complication | during the procedure, and 1 day after the procedure
  Other complications related to the procedure, such as pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Jui-An Lin, Dr., Study Chair — Doctor

IPD SHARING:
Plan to Share IPD: No
There's no plan of sharing individual participant data currently

REFERENCES:
- [Background] Schummer W, Koditz JA, Schelenz C, Reinhart K, Sakka SG. Pre-procedure ultrasound increases the success and safety of central venous catheterizationdagger. Br J Anaesth. 2014 Jul;113(1):122-9. doi: 10.1093/bja/aeu049. Epub 2014 Mar 18. PMID 24648131